CLINICAL TRIAL: NCT00297505
Title: Serotonin, Impulsivity, and Cocaine Dependence Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA008425 (NIH)
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2006-02

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; citalopram; impulsivity; serotonin
MeSH Terms: conditions — Cocaine-Related Disorders; Impulsive Behavior | interventions — Citalopram

INTERVENTIONS:
Drug: citalopram

SUMMARY:
The purpose of this study is to compare the effects of citalopram versus placebo given in the context of contingency management for cocaine dependence.

DETAILED DESCRIPTION:
Cocaine dependence continues to be a significant public health problem, for which there is no FDA approved pharmacotherapy. This study is a 12-week, double blind, placebo controlled trial of citalopram for cocaine dependence. The primary outcome measure is benzoylecgonine positive urines. Secondary measures of side effects and craving are also examined.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects age 18 to 50 who currently meet DSM-IV criteria for cocaine dependence.
* female subjects: a negative pregnancy test

Exclusion Criteria:

* current or past DSM-IV Axis I disorder other than substance abuse/dependence
* any serious non-psychiatric medical illness requiring ongoing medical treatment
* substance dependence other than cocaine within the last 3 months
* negative urine drug screen for cocaine at time of testing
* for female subjects: a positive pregnancy test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2001-04; Study Completion 2004-11

PRIMARY OUTCOMES:
The presence of cocaine metabolites in urine weekly.

SECONDARY OUTCOMES:
Retention rate and cocaine cravings weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas - Houston Health Science Center, Houston, Texas, United States

REFERENCES:
- [Derived] Moeller FG, Schmitz JM, Steinberg JL, Green CM, Reist C, Lai LY, Swann AC, Grabowski J. Citalopram combined with behavioral therapy reduces cocaine use: a double-blind, placebo-controlled trial. Am J Drug Alcohol Abuse. 2007;33(3):367-78. doi: 10.1080/00952990701313686. PMID 17613964